CLINICAL TRIAL: NCT04772287
Title: Adjuvant Toripalimab Versus Placebo Combined With Chemotherapy for EGFR/ALK Mutation Negative Stage II-IIIB(N2) Non-small-cell Lung Cancer (LungMate-008): a Randomised, Double-blind, Controlled, Phase 3 Trial
Brief Title: Adjuvant Toripalimab Plus Chemotherapy for EGFR/ALK Mutation Negative Stage II-IIIB(N2) NSCLC (LungMate-008)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of thoracic department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LungMate-008
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; Cisplatin; Carboplatin; Pemetrexed; Docetaxel; Gemcitabine; Vinorelbine; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab (Experimental)
  Interventions: Drug: Toripalimab
- Placebo (Placebo Comparator)
  Interventions: Drug: Toripalimab mimetic (placebo)

INTERVENTIONS:
Drug: Toripalimab — Toripalimab: 240mg, IV, q3w, 4 cycles in total; Platinum-containing dual-drug chemotherapy: The specific dose is based on the standard of the selected protocol, IV, q3w, a total of 4 cycles.
  Other Names: Cisplatin/Carboplatin; Pemetrexed (non-squamous cell carcinoma)/ Docetaxel/ Gemcitabine/ Vinorelbine/ Paclitaxel
  Arms: Toripalimab
Drug: Toripalimab mimetic (placebo) — Placebo: 240mg, IV, q3w, 4 cycles in total; Platinum-containing dual-drug chemotherapy: The specific dose is based on the standard of the selected protocol, IV, q3w, a total of 4 cycles.
  Other Names: Cisplatin/Carboplatin; Pemetrexed (non-squamous cell carcinoma)/ Docetaxel/ Gemcitabine/ Vinorelbine/ Paclitaxel
  Arms: Placebo

SUMMARY:
This is a randomized, controlled, double-blind, single-center Phase III clinical study in patients with EGFR/ALK mutation negative stage II-IIIB (N2) non-small cell lung cancer (NSCLC) after complete tumor resection. To evaluate the effectiveness and safety of toripalimab compared with placebo combined with platinum-containing dual-drug chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study, understand the research procedures and be able to sign written informed consent.
2. Age ≥18 years old.
3. Histological diagnosis of primary non-small cell lung cancer (NSCLC).
4. An MRI or CT scan of the brain must be performed before lung cancer resection, and it is confirmed that there is no brain metastasis. For patients who have not been examined before surgery, if they have a brain MRI or CT scan before randomization and it is confirmed that there is no brain metastasis, they can still be enrolled.
5. Total resection of primary lung cancer (R0) and systemic lymph node dissection must be performed: complete resection includes lobectomy, sleeve resection, and bilobectomy; systemic lymph node dissection includes hilar and mediastinal lymph node dissection Or sampling, including at least 6 groups of lymph nodes, of which 3 groups are from intrapulmonary (lobar, interlobar or segment) and hilar lymph nodes, and 3 groups are from mediastinal lymph nodes including subcarinal lymph nodes; all surgical margins must be tumor-negative; respectively; The removed mediastinal lymph nodes or the marginal lymph nodes of the removed lung lobes cannot have extranodal invasion.
6. Postoperative pathologically confirmed NSCLC patients with stage II, IIIA and IIIB (N2), the disease is staged according to the American Joint Committee on Cancer (AJCC) 8th edition lung cancer staging standard.
7. Confirmed as negative for EGFR/ALK mutation.
8. Complete recovery from surgery during randomization, and complete postoperative wound healing must be achieved after any surgery;
9. The Eastern Cooperative Oncology Group (ECOG) physical status (PS) score is 0 or 1 and has not deteriorated 2 weeks before the first administration of the study drug, and the minimum expected survival is greater than 12 weeks.
10. Other major organs (liver, kidney, blood system, etc.) function well:

    * Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet ≥100×10^9/L, hemoglobin ≥90 g/L. Note: Patients shall not receive blood transfusion or growth factor support within 14 days before blood collection during the screening period;
    * International normalized ratio (INR) or prothrombin time (PT)≤1.5×upper limit of normal (ULN);
    * Activated partial thromboplastin time (APTT)≤1.5×ULN;
    * Serum total bilirubin≤1.5×ULN (total bilirubin in patients with Gilbert syndrome must be <3×ULN);
    * Aspartic acid and alanine aminotransferase (AST and ALT) ≤2.5×ULN
11. Female patients of childbearing age are willing to take appropriate contraceptive measures (Appendix K) and should not breastfeed from signing informed consent to the end of the study medication within 6 months (whichever occurs later); male patients are effective from signing informed consent Willingness to use barrier contraception (i.e. condoms) within 6 months of the end of sexual evaluation/study medication (whichever occurs later).
12. Female patients have a negative blood pregnancy test result within 7 days before randomization, or meet one of the following criteria to prove that there is no risk of pregnancy:

    1. Postmenopausal is defined as amenorrhea at least 12 months after the age is greater than or equal to 50 years and all exogenous hormone replacement therapy is stopped;
    2. Women younger than 50 years old, if you stop all exogenous hormone treatments and have amenorrhea for 12 months or more, and the levels of luteinizing hormone (LH) and follicle stimulating hormone (FSH) are within the reference range of postmenopausal laboratory Can be considered post-menopausal;
    3. Have received irreversible sterilization, including hysterectomy, bilateral ovarian removal, or bilateral fallopian tube resection, except for bilateral tubal ligation.

Exclusion Criteria:

1. Unresectable or metastatic disease, pathology report showing positive surgical margins or extranodal invasion under the microscope, or leftover lesions during surgery.
2. Patients with lung adenocarcinoma with clear EGFR mutation or ALK rearrangement.
3. Upper sulcus lung cancer.
4. Only patients undergoing segmental resection or wedge resection.
5. Because NSCLC has previously received any anti-cancer treatment other than surgery, including preoperative and postoperative chemotherapy, radiotherapy, targeted therapy (such as small molecule tyrosine kinase inhibitors targeting EGFR, VEGFR and other pathways, monoclonal Antibodies, etc.), immunotherapy, research therapy, etc.; within 14 days before the first administration of the research drug, Chinese medicines and Chinese medicine preparations with anti-tumor therapy indications or tumor adjuvant therapy effects have been used;
6. Suffered from other malignant tumors before the start of the trial, except for the following medical history:

   * Malignant tumors that have been cured, have been inactive for more than 5 years and have a very low risk of recurrence before being selected for the study;
   * Adequately treated non-melanoma skin cancer or malignant lentigines with no evidence of disease recurrence;
   * Carcinoma in situ with adequate treatment and no evidence of disease recurrence;
   * Localized prostate cancer after radical surgery.
7. Complicated with unstable systemic diseases, including active infections, uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg), unstable angina pectoris, attacks that have started within the last 3 months Angina pectoris, congestive heart failure (≥ New York Heart Association [NYHA] level II), myocardial infarction (6 months before enrollment), severe arrhythmia requiring medication, liver, kidney or metabolic diseases;
8. Active, known or suspected autoimmune diseases, or autoimmune paraneoplastic syndromes that require systemic treatment;
9. Subjects who have used corticosteroids (>10 mg/day of prednisone or other equivalent hormones) or other immunosuppressive agents for systemic treatment within 2 weeks before the first administration. In the absence of active autoimmune diseases, inhaled or topical corticosteroids are allowed, and adrenal hormone replacement therapy with a dose of ≤10 mg/day prednisone is allowed;
10. Have significant clinically significant bleeding symptoms or obvious bleeding tendency within 1 month before the first administration, such as gastrointestinal bleeding, gastric ulcer bleeding, active hemoptysis or vasculitis.
11. Arteriovenous thrombosis, such as deep vein thrombosis, pulmonary embolism, etc. occurred within 3 months before the first administration (except for implantable venous port, catheter-derived thrombosis or superficial venous thrombosis, these cases Not considered as "severe" thromboembolism).
12. Diabetic ketoacidosis or hyperglycemia and hyperosmotic state occurred within 6 months before the first administration; fasting blood glucose during the screening period Diabetic patients with ≥7.8 mmol/L or glycosylated hemoglobin test value ≥7.5%.
13. It has been known that there are active infectious diseases, such as active hepatitis B (the virus surface antigen [HBsAg] test result in the screening period is positive and the HBV-DNA test value is ≥2×103 IU/mL) or hepatitis C (defined as the screening period) Hepatitis C virus antibody [HCV-Ab] test result is positive, and HCV-RNA is positive), tuberculosis (there is evidence of active tuberculosis infection within 1 year), syphilis (positive Treponema pallidum specific antibodies and non-specific antibodies), or human immunodeficiency Viral HIV infection (anti-HIV antibody positive), etc.
14. Allergic to test drugs.
15. Previously or currently suffering from interstitial lung disease.
16. Women who are pregnant or breastfeeding.
17. People with neurological diseases or mental illnesses who cannot cooperate.
18. At the same time participate in another therapeutic clinical research.
19. Other situations considered unsuitable by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Estimated)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | up to 40 months
  It refers to the time from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).

SECONDARY OUTCOMES:
Overall survival (OS) | up to 60 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Safety: frequency of severe adverse events | up to 18 months
  The frequency of severe adverse events from the participants enrolling to 90 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.
Health related quality of life (HRQol) | up to 12 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.
5-year overall survival rate | From the completion of the intervention to 5 years.
  Five-year survival rate measures survival at 5 years after treatment.

IPD SHARING:
Plan to Share IPD: Undecided